CLINICAL TRIAL: NCT05215470
Title: CLARA: Characterization of Somatic and Germline Mechanisms That Impact the Immunotherapy Treatment and Prognosis of Patients With Renal Cancer
Brief Title: CLARA: Somatic and Germline Mechanisms That Impact Renal Cancer Immunotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital das Clínicas de Ribeirão Preto (Other)
Collaborators: Bristol-Myers Squibb (Industry); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Leandro M Colli, MD PhD, Head of Oncology, Hospital das Clínicas de Ribeirão Preto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLARA; U1111-1267-7778 (Registry Identifier: UTN - WHO); CA209-6E3 (Other: BMS)
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Renal Cancer Metastatic
Keywords: Renal Cancer; Nivolumab; Ipilimumab; Immunotherapy; molecular profiling
MeSH Terms: conditions — Kidney Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab+Ipilimumab (Experimental): Nivolumab IV 3mg/kg 3/3w + Ipilimumab 1mg/kg 3/3w 4 doses, followed by Nivolumab IV 480mg 4/4w until progression, toxicity, or up to 2 years of use.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is called an anti-PD-1 (Programmed Cell Death Ligand 1) or a checkpoint inhibitor and is an antibody (a type of human protein) designed to allow the body's own immune system to destroy tumors
  Other Names: Opdivo
Drug: Ipilimumab — Ipilimumab is called an anti-CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) and is a type of antibody that works to prevent the body's immune system from stopping to fight a specific cancer
  Other Names: Yervoy

SUMMARY:
The study is studying the joint contribution and interactions of germline variants and somatic mutations and their impact on Renal Cell Carcinoma (RCC) development and treatment (immunotherapy).

DETAILED DESCRIPTION:
One hundred newly diagnosticated stage IV RCC patients will be recruited in the Ribeirao Preto Medical School.

Patients will be treated with immune checkpoint inhibitors (ICI) combination: nivolumab (3 mg/kg of body weight) plus ipilimumab (1 mg/kg) intravenously every three weeks for four doses, followed by nivolumab 480mg every four weeks, until progression, toxicity or complete two years of treatment.

Patients will be followed up for the clinical outcome (progression-free survival, best response, and overall survival).

Fresh-frozen primary tumor tissue will be collected for somatic genomic characterization.

Blood DNA will be genotyped for the identification of common germline variation, as well as ancestry determination.

ELIGIBILITY:
Inclusion Criteria:

* Renal cell carcinoma patient: histological confirmed clear cell tumor;
* First-line metastatic treatment;
* Stage IV with at least one measured lesion;
* Fresh-frozen primary tumor tissue available;
* No previous immunotherapy or tyrosine kinase inhibitor treatment;
* All International Metastatic RCC Database Consortium (IMDC) Risk Score;
* Karnofsky Performance Scale (KPS) >=70;
* >=18 years old.

Exclusion Criteria:

* History of a known or suspected autoimmune disease;
* Any condition requiring systemic treatment with corticosteroids;
* Creatinine clearance < 40mL/min;
* Alanine aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) > 5 x ULN;
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 years
Progression-free survival | 2 years

SECONDARY OUTCOMES:
Overall Response Rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Machado Colli, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirao Preto - USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The research team is committed to sharing data generated by this project with the research community. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to PI.